CLINICAL TRIAL: NCT00265421
Title: The Danish Suture Trial: a Randomized Trial on Perineal Sutures Following Vaginal Birth.
Brief Title: Study of Different Suturing Techniques for Perineal Repair After Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Danish Research Agency (Other); Aase and Ejnar Danielsens Foundation (Other); Aarhus University Hospital (Other); The Danish Midwifery Organization (Unknown); Sophus Jacobsen and wifes´ Foundation (Unknown); Else and Mogens Wedell-Wedellsborgs´ Foundation (Unknown); Frode V. Nyegaard and wifes´ Foundation (Unknown); K. A. Rohde's and wife's Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: The Danish Suture Trial; 2004-70 Etichs Committee
Record Dates: First submitted 2005-12-13; First posted 2005-12-14 (Estimated); Last update posted 2009-09-30 (Estimated); Status verified 2009-09

CONDITIONS: Perineal Lacerations; Episiotomy
Keywords: Suture Techniques
MeSH Terms: interventions — Suture Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Suture technique for perineal repair after delivery

SUMMARY:
We wish to determine wich of two standardized suturing techniques is the best for perineal repair if a perineal laceration or an episiotomy is present after vaginal birth.

The participants are healthy primi para and deliver at term.

DETAILED DESCRIPTION:
A randomised controlled trial with 400 participants was initiated in August 2004. The two suture techniques compared were both 2-layered and either continuous sutures or interrupted, inverted stitches to perineal muscles and the subcuticular layer. A polyglactin 910 multifilament thread on an atraumatic needle was used and the perineal skin was left unsutured. Healthy primiparas >36+0 weeks gestation could participate if they had a either a 2nd degree perineal laceration or an episiotomy.

The trial was a double-blind and analysis was done on an intention-to-treat basis. Main outcomes were pain, wound healing and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

Primipara, 2nd degree perineal laceration or episiotomy. Vaginal birth of one child in occipital position terminating a pregnancy at 36 weeks or later. A soft cup used to deliver the baby was accepted. Participants must be able to understand and speak Danish.

Exclusion Criteria:

Perineal 3rd or 4th degree injuries, post partum haemorrhage extending 1000 ml. or manual removal of placenta, former perineal wounds, foetus mortuus or delivery of a child immediately transferred to the neonatal ward, Diabetes Mellitus, instrumental delivery, Caesarean Section or gemelli.

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 400
Dates: Start 2004-08; Study Completion 2006-04

PRIMARY OUTCOMES:
Pain in perineal area day 1 and 10 after delivery.
Healing of wound day 1 and 10 after delivery.

SECONDARY OUTCOMES:
Patient satisfaction with perineal sutures performed at birth.
Incontinence.
Need for resuturing of perineal area within 1 year after delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Niels Uldbjerg, Professor, Study Chair — Aarhus University Hopspital, dept. of Obst. & Gyn.
Locations (1):
- Dept. of Obstetrics and Gynaecology, Skejby Sygehus, Aarhus, Denmark